CLINICAL TRIAL: NCT00002304
Title: A Randomized Comparative Multicenter Trial of Fluconazole and Ketoconazole in the Treatment of Esophageal Candidiasis in Immunocompromised Patients
Brief Title: A Comparison of Fluconazole and Ketoconazole in the Treatment of Fungal Infections of the Throat in Patients With Weakened Immune Systems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pfizer (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 012B; 056-150
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1990-02

CONDITIONS: Candidiasis, Esophageal; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Immune Tolerance; Ketoconazole; Esophagitis; Fluconazole; Acquired Immunodeficiency Syndrome; Candidiasis, Oral
MeSH Terms: conditions — Candidiasis; HIV Infections; AIDS-Related Opportunistic Infections; Esophagitis; Acquired Immunodeficiency Syndrome; Candidiasis, Oral | interventions — Ketoconazole; Fluconazole

INTERVENTIONS:
Drug: Ketoconazole
Drug: Fluconazole

SUMMARY:
To compare the safety, tolerance, and effectiveness of fluconazole and ketoconazole in the treatment of candidal esophagitis in immunocompromised patients.

ELIGIBILITY:
Inclusion Criteria

Prior Medication:

Allowed:

* Cyclosporin if levels can be monitored for proper cyclosporin dose adjustment.

Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Evidence of noncandidal systemic fungal infections.
* Leukopenia (white blood cell count less than 1000/mm3), or expected to develop leukopenia during the study.
* Other condition known to be associated with poor ketoconazole absorption, e.g., hypochlorhydria.
* Leukemia requiring chemotherapy.
* Any other condition which in the opinion of the investigator would make the patient unsuitable for enrollment.

Concurrent Medication:

Excluded:

* Warfarin.
* Immunostimulants.
* Interferon.
* Oral or topical antifungal agents.

Concurrent Treatment:

Excluded:

* Lymphocyte replacement.

Patients with the following are excluded:

* History of allergy to imidazoles.
* Abnormalities which may preclude esophagoscopy or endoscopy before or during the study.
* Inability to tolerate fluconazole or ketoconazole.
* Inability or unwillingness to give written informed consent.
* Life expectancy < 2 months.

Prior Medication:

Excluded:

* Rifampin or ansamycin, pending clarification of drug interactions between these drugs and fluconazole.
* Warfarin.

Patients must meet the CDC criteria for the diagnosis of AIDS or be otherwise immunocompromised (e.g., malignancy, renal transplant) and have a diagnosis of oral candidiasis and/or esophageal symptoms of dysphagia and/or odynophagia.

Illicit or illegal drug use.

Ages: 13 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (42):
- United States (41):
  - Good Samaritan Med Ctr, Phoenix, Arizona
  - Arkansas Children's Hosp, Little Rock, Arkansas
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - Eisenhower Med Ctr, Rancho Mirage, California
  - ViRx Inc, San Francisco, California
  - UCSF Hosp, San Francisco, California
  - George Washington Univ Med Ctr, Washington D.C., District of Columbia
  - Regional Oncology Ctr, Daytona Beach, Florida
  - Ctr for Special Immunology, Fort Lauderdale, Florida
  - Mem Hosp Hollywood, Hollywood, Florida
  - Med Ctr Clinic, Pensacola, Florida
  - St Petersburg Med Clinics, St. Petersburg, Florida
  - Georgia Baptist Med Ctr, Atlanta, Georgia
  - DeKalb Gen Hosp, Decatur, Georgia
  - Gwinnett Med Ctr, Lawrenceville, Georgia
  - Atlanta Hosp, Riverdale, Georgia
  - Clayton Gen Hosp, Riverdale, Georgia
  - Dr Winkler Weinberg, Roswell, Georgia
  - Univ Hosp, Boston, Massachusetts
  - Baystate Med Ctr of Springfield, Springfield, Massachusetts
  - Leila Hosp and Health Care Ctr, Battle Creek, Michigan
  - Harper Hosp, Detroit, Michigan
  - Butterworth Hosp, Grand Rapids, Michigan
  - Holland Community Hosp, Holland, Michigan
  - Munson Med Ctr, Traverse City, Michigan
  - Dr Eugene Speck, Las Vegas, Nevada
  - Univ of New Mexico School of Medicine, Albuquerque, New Mexico
  - SUNY / Health Sciences Ctr at Brooklyn, Brooklyn, New York
  - Roswell Park Memorial Institute, Buffalo, New York
  - Cornell Univ Med Ctr, New York, New York
  - Bowman Gray School of Medicine / North Carolina Baptist Hosp, Winston-Salem, North Carolina
  - Buckley Braffman Stern Med Associates, Philadelphia, Pennsylvania
  - Wilson Brailsford Clinic, Spartanburg, South Carolina
  - Baroness Erlanger Hosp, Chattanooga, Tennessee
  - Univ of Tennessee, Memphis, Tennessee
  - Univ TX Galveston Med Branch, Galveston, Texas
  - Audie L Murphy Veterans Administration Hosp, San Antonio, Texas
  - Univ TX San Antonio Health Science Ctr, San Antonio, Texas
  - Infectious Disease Physicians Inc, Annandale, Virginia
  - McGuire Virginia Med Ctr, Richmond, Virginia
  - Virginia Mason Med Ctr, Seattle, Washington
- Henderson Gen Hosp, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Laine L, Dretler RH, Conteas CN, Tuazon C, Koster FM, Sattler F, Squires K, Islam MZ. Fluconazole compared with ketoconazole for the treatment of Candida esophagitis in AIDS. A randomized trial. Ann Intern Med. 1992 Oct 15;117(8):655-60. doi: 10.7326/0003-4819-117-8-655. PMID 1308663